CLINICAL TRIAL: NCT00386230
Title: Short ZDV Course to Prevent Perinatal HIV in Thailand
Brief Title: Shortened Zidovudine Regimens to Prevent Mother-to-Child Transmission of HIV Type 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut de Recherche pour le Developpement (Other Government)
Collaborators: Harvard School of Public Health (HSPH) (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PHPT-1; NIH 5 R01 HD33326-05
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2008-05-02 (Estimated); Status verified 2008-05

CONDITIONS: HIV Infections; Pregnancy
Keywords: transmission; infant; HIV; pregnancy; HIV-1 infection; HIV Seronegativity
MeSH Terms: conditions — HIV Infections

ARMS (4):
- 1 (Experimental): Maternal ZDV treatment starting at 35 weeks Gestational Age (GA) and continuing through labor and delivery, and three days of infant ZDV treatment starting at birth (Smother-Sinfant)
  Interventions: Drug: ZDV Short (mother)-Short (infant): Comparison of zidovudine durations
- 2 (Experimental): Maternal ZDV treatment starting at 35 weeks Gestational Age (GA) and continuing through labor and delivery, and six weeks of infant ZDV treatment starting at birth (Smother-Linfant)
  Interventions: Drug: ZDV Short (mother)-Long (infant): Comparison of zidovudine durations
- 3 (Experimental): Maternal ZDV treatment starting at 28 weeks Gestational Age (GA) and continuing through labor and delivery, and three days of infant ZDV treatment starting at birth (Lmother-Sinfant)
  Interventions: Drug: ZDV Long (mother)-Short (infant): Comparison of zidovudine durations
- 4 (Active Comparator): Maternal ZDV treatment starting at 28 weeks Gestational Age (GA) and continuing through labor and delivery, and six weeks of infant ZDV treatment starting at birth (Lmother-Linfant). This study arm was the reference regimen.
  Interventions: Drug: ZDV Long (mother)-Long (infant): Comparison of zidovudine durations

INTERVENTIONS:
Drug: ZDV Short (mother)-Short (infant): Comparison of zidovudine durations — Maternal ZDV treatment (300 mg, twice daily) starting at 35 weeks Gestational Age (GA) until the onset of labor, ZDV 300 mg at the onset of labor and then 300 mg every 3 hours until delivery. Three days of infant ZDV treatment (2 mg/kg, every 6 hours) starting at birth (Smother-Sinfant)
  Arms: 1
Drug: ZDV Short (mother)-Long (infant): Comparison of zidovudine durations — Maternal ZDV treatment (300 mg, twice daily) starting at 35 weeks Gestational Age (GA) until the onset of labor, ZDV 300 mg at the onset of labor and then 300 mg every 3 hours until delivery. Six weeks of infant ZDV treatment (2 mg/kg, every 6 hours) starting at birth (Smother-Linfant)
  Arms: 2
Drug: ZDV Long (mother)-Short (infant): Comparison of zidovudine durations — Maternal ZDV treatment (300 mg, twice daily) starting at 28 weeks Gestational Age (GA) until the onset of labor, ZDV 300 mg at the onset of labor and then 300 mg every 3 hours until delivery. Three days of infant ZDV treatment (2 mg/kg, every 6 hours) starting at birth (Lmother-Sinfant)
  Arms: 3
Drug: ZDV Long (mother)-Long (infant): Comparison of zidovudine durations — Maternal ZDV treatment (300 mg, twice daily) starting at 28 weeks Gestational Age (GA) until the onset of labor, ZDV 300 mg at the onset of labor and then 300 mg every 3 hours until delivery. Six weeks of infant ZDV treatment (2 mg/kg, every 6 hours) starting at birth (Lmother-Linfant)
  Arms: 4

SUMMARY:
The purpose of the study was to test the equivalence of a short zidovudine (ZDV) regimen as compared to a longer, ACTG-076-like, ZDV regimen in reducing the risk of mother-to-child transmission of HIV: and to assess and compare the safety and tolerance of the long and shortened ZDV regimens.

DETAILED DESCRIPTION:
Multicenter, randomized, four arms, double-blind, controlled study. Consenting pregnant women were tested for HIV from the beginning of pregnancy until 26 of gestational age (GA). If HIV-positive and eligible, women completed a Pre-entry baseline check-up. Enrollment took place at 28 weeks' gestational age. Women meeting selection criteria were randomly assigned to one of four study arms (see below).

AMENDMENT (March 20, 1999)

Data Safety and Monitory Board interim review (March 17, 1999) The DSMB reported that the transmission rate in the longest arm (long treatment of both mother and baby), was significantly lower than that in the shortest arm (short treatment of both the mother and the baby) and this discrepancy was larger than the previously agreed on difference which, if found, would call for changing the study design. In addition, the transmission rates in the remaining two arms of the study were similar to that in the longest arm. The difference that was found could not be explained by any baseline characteristics of the participants, such as maternal age, gestational age at delivery, birth weight, cesarean section rate, or any others.

The DSMB recommended that enrollment into the shortest arm of the study be terminated, and the study be continued with a modification of design so that new enrollees would enter one of the three remaining arms.

All women enrolled before this amendment was effective and delivering after March 20th, 1999, and previously randomized to the Smother-Sinfant arm, were unblinded in order to give their infants open label zidovudine for 6 weeks.

ELIGIBILITY:
Pre-inclusion

Women are eligible for Pre-Entry if they:

* have evidence of HIV infection (confirmed on a second sample);
* present themselves for prenatal care before 26 weeks GA, based on last menstrual period and/or sonogram results;
* intend to stay in the province for at least 18 months after delivery;
* can provide informed consent;
* have given written informed consent to participate in the study;
* intend to carry the pregnancy to term.

Inclusion Criteria:

* all pre-entry criteria;
* date of enrollment: 28 weeks GA, based on last menstrual period and/or sonogram results;
* the following laboratory values within 21 days prior to randomization:
* hemoglobin > 8.0 g/dL;
* absolute neutrophil count > 750 cells/mm3;
* SGPT < 5 x upper limit of normal;
* serum creatinine < 1.5 mg/dL (women with a serum creatinine > 1.5 mg/dL must have a measured eight-hour urine creatinine clearance > 70 mL/min.);
* agreement not to breastfeed.

Exclusion Criteria:

* AIDS according to the Thai Communicable Diseases Control (CDC) classification;
* pre-existing maternal/fetal condition that contraindicates the use of ZDV
* oligohydramnios, unexplained polyhydramnios, fetal hydrops or ascites or other evidence of pre-existing in-utero anemia;
* clinically significant history of intolerance to ZDV treatment resulting in discontinuation of therapy for more than 4 weeks;
* receipt of ZDV during the current pregnancy for any indication, or women who need ZDV for their own health (women are then followed separately);
* receipt of other antiretroviral agents, passive immunotherapy, anti-HIV vaccines, cytolytic agents (usually referred as chemotherapy), radiation therapy, or corticosteroids during this pregnancy except steroids less than 7 (see Zidovudine Investigator's Brochure);
* simultaneous participation in another clinical trial.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1554
Dates: Start 1997-06; Study Completion 2000-08 (Actual)

PRIMARY OUTCOMES:
Definitive HIV infection in children as assessed by positive PCR on two peripheral blood samples collected at two separate occasions.

SECONDARY OUTCOMES:
Safety: clinical and biological assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Lallemant, MD, Principal Investigator — Institut de Recherche pour le Developpement
Locations (1):
- Phpt - Ird 174, Chiang Mai, Chiang Mai, Thailand

REFERENCES:
- [Result] Lallemant M, Jourdain G, Le Coeur S, Kim S, Koetsawang S, Comeau AM, Phoolcharoen W, Essex M, McIntosh K, Vithayasai V. A trial of shortened zidovudine regimens to prevent mother-to-child transmission of human immunodeficiency virus type 1. Perinatal HIV Prevention Trial (Thailand) Investigators. N Engl J Med. 2000 Oct 5;343(14):982-91. doi: 10.1056/NEJM200010053431401. PMID 11018164
- [Derived] Sripan P, Le Coeur S, Amzal B, Ingsrisawang L, Traisathit P, Ngo-Giang-Huong N, McIntosh K, Cressey TR, Sangsawang S, Rawangban B, Kanjanavikai P, Treluyer JM, Jourdain G, Lallemant M, Urien S. Modeling of In-Utero and Intra-Partum Transmissions to Evaluate the Efficacy of Interventions for the Prevention of Perinatal HIV. PLoS One. 2015 May 19;10(5):e0126647. doi: 10.1371/journal.pone.0126647. eCollection 2015. Erratum In: PLoS One. 2015 Jun 26;10(6):e0130917. doi: 10.1371/journal.pone.0130917. PLoS One. 2015 Aug 28;10(8):e0137368. doi: 10.1371/journal.pone.0137368. PMID 25992639